CLINICAL TRIAL: NCT01771913
Title: Immunophenotyping of Fresh Stromal Vascular Fraction From Adipose Derived Stem Cells (ADSC) Enriched Fat Grafts for Refinements of Reconstructed Breasts
Brief Title: Immunophenotyping of Fresh Stromal Vascular Fraction From Adipose Derived Stem Cells (ADSC) Enriched Fat Grafts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luiz Alexandre Lorico Tissiani, MD, Chief of Breast Reconstructive Unit at Hospital Municipal Carmino Caricchio, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: boosteredADSCs
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-07

CONDITIONS: Breast Reconstruction; Contour Irregularities; Volume Insufficiency
Keywords: adipocytes; cell transplantations; mesenchymal stem cell; immunophenotyping; adipose tissue; breast reconstruction; mammaplasty; magnetic resonance imaging; fat necrosis
MeSH Terms: conditions — Fat Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- centrifuged fat graft (Sham Comparator): female patients who underwent breast reconstruction and present with volume insufficiency will undergo centrifuged fat graft for contour and volume refinements.
  Interventions: Genetic: centrifuged fat graft
- ADSCs enriched centrifuged fat graft (Active Comparator): female patients who underwent breast reconstruction and present volume insufficiency will undergo ADSCs enriched fat grafting for volume and irregularity contour improvement
  Interventions: Genetic: ADSCs enriched fat graft

INTERVENTIONS:
Genetic: centrifuged fat graft — fat from the abdominal subcutaneous tissue will be taken by vacuum assisted lipectomy and immediately prepared to be grafted in the reconstructed breast that presents contour irregularities and/or volume insufficiency. No adipose derived stem cells will enrich the fat grafts in this group.
  Arms: centrifuged fat graft
Genetic: ADSCs enriched fat graft — fat from the abdominal subcutaneous tissue will be taken by suction assisted lipectomy and stromal vascular fraction will be isolated and immediately added to the fat graft that will be employed to improve contour irregularities and volume insufficiency of reconstructed breasts.
  Arms: ADSCs enriched centrifuged fat graft

SUMMARY:
The purpose of this study is to investigate if there is a relationship between the take of fat grafts with and without ADSCs and the presence of specific surface markers on the cells of the stromal vascular fraction.

DETAILED DESCRIPTION:
Two groups of patients will be studied. The control will receive centrifuged fat grafts while the other group will receive centrifuged enriched fat grafts with ADSCs. The performance of both grafts will be assessed through volume measurement employing MRI before and after 6 months post-op.

ELIGIBILITY:
Inclusion Criteria:

* contour irregularities and volume insufficiency in reconstructed breasts no matter the method of reconstruction employed
* local flaps with conditions to receive fat grafts
* good health condition

Exclusion Criteria:

* breast cancer patients under chemotherapy
* smokers
* bad health condition
* patients too thin
* patients that require a new reconstructive surgery (secondary reconstruction)

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nivaldo Alonso, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Hospital Municipal Carmino Caricchio, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Spear SL, Wilson HB, Lockwood MD. Fat injection to correct contour deformities in the reconstructed breast. Plast Reconstr Surg. 2005 Oct;116(5):1300-5. doi: 10.1097/01.prs.0000181509.67319.cf. PMID 16217471
- [Result] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Result] Gimble JM, Bunnell BA, Casteilla L, Jung JS, Yoshimura K. Phases I-III Clinical Trials Using Adult Stem Cells. Stem Cells Int. 2011 Feb 23;2010:604713. doi: 10.4061/2010/604713. No abstract available. PMID 21461337
- [Result] Yoshimura K, Sato K, Aoi N, Kurita M, Hirohi T, Harii K. Cell-assisted lipotransfer for cosmetic breast augmentation: supportive use of adipose-derived stem/stromal cells. Aesthetic Plast Surg. 2008 Jan;32(1):48-55; discussion 56-7. doi: 10.1007/s00266-007-9019-4. Epub 2007 Sep 1. PMID 17763894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients who have contour irregularities after any method of breast reconstruction. recruited from jan/2012 to august/2014.
Period: Overall Study
Arm/Group | Centrifuged Fat Graft | ADSCs Enriched Centrifuged Fat Graft
Started | 9 | 11
Completed | 8 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Centrifuged Fat Graft | ADSCs Enriched Centrifuged Fat Graft | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 11 | 18
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.5) | 49.6 (5.7) | 49.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 8 | 11 | 19
breast volume [Mean (Standard Deviation); unit: mL] | 562.8 (187.7) | 650.1 (206.8) | 613.3 (198.5)

OUTCOME MEASURES:

1. Primary Outcome: Volume Maintenance
Description: Volumetry of the reconstructed breasts will be accomplished through MRI and OsiriX software. Osirix software allows breast volume calculation through the determination of regions of interest (ROIs) on an MRI sequence. Once the pre (V1) and postoperative (V2) volumes were determined the following formula was applied: (V2 - V1) X 100/graft volume. The result, expressed in percentage, expresses graft volume persistence.
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: percentage of graft volume persistency
Arm/Group | Centrifuged Fat Graft | ADSCs Enriched Centrifuged Fat Graft
Number analyzed (Participants) | 8 | 11
percentage of graft volume persistency | 51.6 (18.4) | 78.9 (74.9)
Statistical Analysis 1: Comparison: Centrifuged Fat Graft vs ADSCs Enriched Centrifuged Fat Graft; Test type: Superiority or Other; p = 0.310, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Immunophenotyping
Description: Immunophenotyping of the fresh stromal vascular fraction of both groups. Immunophenotyping or flow cytometry measures how many cells, in a sample, express a specific surface marker. A surface marker or a group of markers may characterize a specific cell type. The software that accompanies the flow cytometer determines the number of cells (in percentage) that express the tested surface marker.
Time Frame: baseline
Population: we had technical problems in processing 4 tissue samples in each arm.
Measure: Mean (Standard Deviation); unit: percentage of expression for CD90
Arm/Group | Centrifuged Fat Graft | ADSCs Enriched Centrifuged Fat Graft
Number analyzed (Participants) | 4 | 7
percentage of expression for CD90 | 27 (27.9) | 79 (15.4)
Statistical Analysis 1: Comparison: Centrifuged Fat Graft vs ADSCs Enriched Centrifuged Fat Graft; Test type: Superiority or Other; p = 0.026, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Number of Participants Experiencing Fat Necrosis in the Postoperative Period
Description: Fat necrosis may occur whenever a fat graft is performed and it has clinical relevance. It can emerge as oil cysts or small nodules a little bit painful. In mammograms of normal breasts, fat necrosis present as cysts or micro calcifications that present a benign appearance. In breast reconstruction patients, fat necrosis, despite its benign characteristics, can suggest cancer recurrence.
Time Frame: up to 3 years
Measure: Number; unit: participants
Arm/Group | Centrifuged Fat Graft | ADSCs Enriched Centrifuged Fat Graft
Number analyzed (Participants) | 8 | 11
participants | 0 | 4
Statistical Analysis 1: Comparison: Centrifuged Fat Graft vs ADSCs Enriched Centrifuged Fat Graft; Test type: Superiority or Other; p = 0.103, Fisher Exact

ADVERSE EVENTS:
Time Frame: from fat grafting to 3 years (average) for ADSC arm and 16 months for the centrifuged arm.
Arm/Group | Centrifuged Fat Graft | ADSCs Enriched Centrifuged Fat Graft
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No